CLINICAL TRIAL: NCT05646953
Title: A Proof-of-Concept, Safety and Efficacy Study of Vasu Facial Beauty Oil in Healthy Adult Human Subjects
Brief Title: Safety and Efficacy Study of Vasu Facial Beauty Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Vasu Healthcare Private Limited (Industry)
Responsible Party: Principal Investigator, Dr Nayan Patel, Medical Director, NovoBliss Research Pvt Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB220033-VH
Record Dates: First submitted 2022-12-03; First posted 2022-12-12 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Healthy; Wrinkle; Dry Skin; Skin Pigment
Keywords: Healthy, Dry Skin, Wrinkles, Pigmentation, Safety, Efficacy
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Intervention Model Description: Single Center, Open Label, Safety and Efficacy
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vasu Facial Beauty Oil (Experimental): Vasu Facial Beauty Oil blends the Traditional Beauty recipe of Kumkumadi Tailam with clinically- proven Natural Plant Actives to offer a unique product that gives a Natural Glow to face, overcoming hyper-pigmentation, age spots, wrinkles, and blemishes with Avacado, Lavender, Argan, Rapeseed.
  Kumkumadi Oil is an Ayurvedic Elixir that is effective for many skincare concerns such as Hyperpigmentation, Dark spots, Age spots, Acne scars, Fine lines, Wrinkles as well as Dark circles. It is also used for Beautifying, Rejuvenating and Uplifting the skin.
  Interventions: Other: Facial Beauty Oil

INTERVENTIONS:
Other: Facial Beauty Oil — Mode of Usage Step 1- Wash face, pat dry Step 2 - Gently massage 2-3 drops of Vasu Facial Beauty Oil over the face and neck till it gets absorbed and keep it overnight.
  Step 3 - Use it for 60 days Frequency - Daily before going to bed. Route of Administration - Topical
  Other Names: Vasu Facial Beauty Oil

SUMMARY:
This is an open-label, single-arm, single-center, proof-of-concept, exploratory, safety and efficacy, clinical study of a Vasu Facial Beauty Oil in healthy adult human subjects.

Considering the proof of concept study, a sufficient number [maximum of 32 subjects (25 females and 7 males)] of adult subjects will be recruited/enrolled to ensure a total of 30 subjects complete the study.

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. The total clinical study duration is 60 Days from Day 01.

DETAILED DESCRIPTION:
This is an open-label, single-arm, single-center, proof-of-concept, exploratory, safety and efficacy, clinical study of a Vasu Facial Beauty Oil in healthy adult human subjects.

Considering proof of concept study, a sufficient number [maximum of 32 subjects (25 females and 7 males)] of adult subjects will be recruited/enrolled to ensure a total of 30 subjects complete the study.

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. The adult female/male subjects will be instructed to visit the facility as per the below visits.

* Visit 01 (Day 01): Screening, Enrolment, Baseline Evaluations
* Visit 02 (Day 30 i.e. week 4): Treatment Period, Evaluations
* Visit 03 (Day 60 i.e. week 8): Evaluations, End of Study Visit Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called on the telephone by the recruiting department prior to the enrolment visit. Subjects will be told during screening (prior to enrolment) not to wear any facial make-up or use any hair product on the study visit day.

Assessment of efficacy parameters before test product usage will be done on day 1, and after test, product usage will be done on day 30, and day 60 as listed below.

* Skin Elasticity: Derma Lab Combo or Cutometer Dual MPA 580 (Right Cheek)
* MoistureMeterEPiD: Skin Hydration (Right cheek)
* Vapometer: Skin Barrier function - Transepidermal water loss (Right cheek)
* Skin Colorimeter CL 400: Right cheek skin colour evenness L*, a* b*, ITA Angle (Individual Typology Angle)
* Visioscan: Crow's feet area wrinkles, fine lines, skin texture - roughness, dryness, wrinkles, smoothness
* Physician Global Assessments (PGA) scoring using Griffiths scale - Skin dryness, redness, fine wrinkling/lines, coarse wrinkling/lines, laxity, roughness, and sallowness
* Glogau Skin Age
* Skin Pigmentation Scoring
* Occurrence of Acne - Investigator Global Assessment (IGA) score for assessment of Acne Severity
* Digital Photographs: Facial photographs Before test product usage and after test product usage using DermoPrime or equivalent.
* Subjective Product Perception Assessment regarding the test product's effect on skin firmness, appearance, radiance, the occurrence of acne breakouts, glowing skin tone, blemishes, dark skin patch removal, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 25 to 55 years (both inclusive) at the time of consent.
2. Sex: Healthy males and non-pregnant/non-lactating females.
3. Females of childbearing potential must have a self-reported negative pregnancy test.
4. Subjects are generally in good health.
5. Subject has a score of at least "mild skin aging" based on Physican Global Assessment (PGA) at screening visit.
6. Subject with Glogau Skin Age II or III as assessed by the Dermatologist/Dermatologist Trained Evaluator.
7. Subjects with wrinkles at Crow's feet area.
8. Subjects with uneven texture skin, uneven skin tone, with dry to normal skin only.
9. Subjects with dry skin having ≤ 40% value as evaluated by MoisturemeterEpiD.
10. Subject is willing to forgo cosmetic procedures 3 months prior to and for the duration of the study.
11. Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
12. Subject is able to follow their normal skin care routines and to refrain from introducing any new skin care products during the study.
13. Subject is able to forgo changes in baseline medications and nutritional supplements during the study period.
14. If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (Intrauterine Device, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
15. If currently using hormonal contraception, has been using this form of contraception for at least 6 months and agrees to continue using the same contraception for the duration of the study.
16. Subjects are willing not to introduce any new soaps, cleansers, laundry detergents, lotions, creams, shampoos etc. for the duration of the study.
17. Subjects are willing to give written informed consent and are willing to follow the study procedure.
18. Subjects who have used other marketed products for hair thinning in the past.
19. Subjects who commit not to use medicated/ prescription shampoos/hair care products (containing Minoxidil / Anti-thinning agents) or any other hair growth, treatment for thin hair, or hair products other than the test product for the entire duration of the study.
20. Willing to use test product throughout the study period.

Exclusion Criteria:

1. Subject has a history of allergy or sensitivity to the test treatment ingredients like Kumkumadi tailam, avocado, argan, lavender, rapeseed oil and others etc.
2. Subject has used any systemic therapy with chronic antibiotic therapy, retinoids, and/or oral steroids during the 4 weeks prior to the start or anticipates having to use at any point during the study.
3. Subject has applied any topical retinoids within 2 weeks of the screening visit or anticipates having to use at any point during the study.
4. Subject is not willing to avoid the unprotected sun or other UV radiation exposure during the study period.
5. Subject is currently pregnant/breastfeeding.
6. Subject has a history of alcohol or drug addiction.
7. Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.
8. Pregnant or breastfeeding or planning to become pregnant during the study period.
9. History of chronic illness which may influence the cutaneous state.
10. Subjects participating in other similar cosmetics, devices or therapeutic trials or skin care products within the last four weeks.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Assessment of Reduction in Facial Wrinkles and Fine lines of Crow's feet area | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  To evaluate the effectiveness of the test product in reducing the facial wrinkles and fine lines of Crow's feet area in healthy adult human subjects using VisioScan (Instrumental Readings).

SECONDARY OUTCOMES:
Physician Global Assessments (PGA) scoring using Griffiths scale - Skin dryness, redness, fine wrinkling/lines, coarse wrinkling/lines, laxity, roughness and sallowness | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  To assess the effect of the test product in terms of change in Physician Global Assessments (PGA) scoring using Griffiths scale - Skin dryness, redness, fine wrinkling/lines, coarse wrinkling/lines, laxity, roughness and sallowness by Dermatologist Trained Evaluator
Assessment of Glogau Skin Age | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  To assess the effect of the test product in terms of change in Glogau Skin Age by Dermatologist Trained Evaluator
Assessment of Skin Pigmentation | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  To assess the effect of the test product in terms of instant change in skin pigmentation by a Dermatologist Trained Evaluator
Assessment of Skin Color L-, a-,b- and ITA (Individual Topology Angle) | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  To assess the effect of the test product in terms of change in skin colour i.e. L* a* b* and ITA (Individual Topology Angle) using Skin-Colorimeter CL 400
Assessment of Facial Skin Elasticity | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  To assess the effect of the test product in improvement in Skin elasticity by DermaLab Combo or Cutometer Dual MPA 580
Assessment in improvement in Skin Hydration | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  To assess the effect of the test product in improvement in Skin hydration by MoistureMeterEPiD
Assessment in improvement in Skin Barrier Function - Transepidermal Water Loss (TEWL) | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  To assess the effect of the test product on improvement in Skin barrier function in terms of decrease in Transepidermal Water Loss (TEWL) using Vapometer
Measurement of Skin Brightness and Skin Pigmentation | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  To assess the effect of test product in terms of change in Skin brightness and skin pigmentation reduction by Dermatologist Trained Evaluator
Assessment of Occurrence of Acne Lesions by Investigator Global Assessment (IGA) scoring | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  To assess the occurrence of Acne lesion in terms of IGA Scoring for Acne Severity by Dermatologist Trained Evaluator
Change in Facial Photograph | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  Change in photograph from "before test product usage" and "after test product usage" using DermoPrime Skin | Hair Analyzer or Equivalent
Assessment of Product Perception - Sensory Attributes | On Day 1 before product usage, on Day 30 and Day 60 after test product usage
  To assess the effect of the test product in terms of treatment perception regarding the test product's effect on skin firmness, appearance, radiance, the occurrence of acne breakouts, glowing skin tone, blemishes, dark skin patch removal, etc. based on study participants subjective ratings

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nayan K Patel, MBBS, Principal Investigator — Medical Director
Locations (1):
- NovoBliss Research Private Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No